CLINICAL TRIAL: NCT04017949
Title: Viscosupplementation and Corticosteroid Knee Injections: Do They Offer Any Benefit in Improving Osteoarthritic Knee Pain
Brief Title: Do Knee Injections Offer Benefit With Knee Arthritis Pain
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, William Vascik, Senior Physician Assistant, University of Pittsburgh
Other Study IDs: STUDY19050002
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Knee Osteoarthritis
Keywords: viscosupplementation injection; corticosteroid injection
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Corticosteroid injection — 1 cc (40 mg) of a corticosteroid (kenalog) is given

SUMMARY:
Corticosteroid and viscosupplementation injections have been used for years to treat osteoarthritic pain in knees. Recent studies have varied in reporting the effectiveness with these injections. None have been found to analyze pain scores between the groups though.

This study aims to evaluate the effectiveness of corticosteroid injection (a single injection of 1 cc of 40 mg kenalog: 4 cc 0.5% Naropin) and viscosupplementation injection (Euflexxa and Synvisc, both are 2 cc of the medication given in 3 injections over a 3 week period). This will be analyzed with a modified visual analog scale over a period of time. An initial VAS will be collected prior to the first injection in the clinic. With the viscosupplementation injections, a VAS will be collected prior to injections 2 and 3 as well. These VAS are logged in the patient's chart. For both types of injections, the participant will be called and a VAS will be recorded 6 weeks post injection and 3 month post injection. These VAS will NOT be logged in the participant's chart. All VAS will be collected/recorded by the principal investigator. Statistical analysis will be conducted with a paired t-test (p<0.05 with a confidence interval at 95%) from the pre-injection VAS and VAS subsequently.

DETAILED DESCRIPTION:
Corticosteroid injections and viscosupplementation (Euflexxa and Synvisc)injections are routine treatments patients receive for knee osteoarthritis. However, studies are limited/flawed outlining their effectiveness. This study aims to analyze the effectiveness of these injections on participant's perception of pain. This will be assessed using a visual analog scale (VAS). VAS scores will be logged pre-injection by the principal investigator. For viscosupplementation injections, a VAS will be logged pre-injection at the second and third office visit. Because there is not immediate improvement with injections a VAS will be logged via phone call 6 weeks post-injection. To assess the long-term effectiveness, a VAS will be logged 3 months post-injection as well.

Participants will be recruited at their office visit scheduled with the principal investigator. Prior to the office visit, one of the surgeons diagnosed the potential participant with knee osteoarthritis. They recommended proceeding with a particular knee injection based upon previous treatments and insurance authorization. The determination of which injection is administered is not being determined by the study need.

The participant will be assigned a number at random at the first visit. The participant will rate their current pain based on the VAS. For participants who receive bilateral injections, they will provide a VAS for each knee. This will be documented prior to administration of the first, second, and third viscosupplementation injection. Because viscosupplementation injections can take up to 6 weeks to be beneficial, a subsequent VAS score will be assessed over the phone by the principal investigator. Because some research suggests a maximum injection benefit of about 14 weeks, the last VAS will be logged at the 3 month period also over the phone, resulting in 5 VAS for each participant. For cortisone injections, an initial VAS will be assessed prior to the injection, followed by a VAS at 6 weeks and 3 months over the phone.

Paired t-test (p<0.05 and confidence interval at 95%) for the pre-injection VAS score and each documented VAS will be analyzed Based upon 2018 statistics, the principal investigator averaged 101 patients per month who received knee injections. The goal is to have a 3 month sample (~300 potential participants). With a CI of 95%, the sample size would need to be 169 participants.

With the looming changes with UPMC/Highmark patient enrollment, the number of Synvisc patients may be reduced. In the event that after the 3 month trial has ended, and there is an inadequate number of subjects who received Synvisc, Synvisc will not included in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* The participant has been previously been diagnosed with knee osteoarthritis by one of the investigator's surgeons in the office.
* The injection was recommended by another clinician
* Age of the pool of participants will be 40 years old and over
* All gender and BMI will be considered
* Severity of osteoarthritis will not be a determinant

Exclusion Criteria:

* Patients who are receiving any injections based upon medical recommendation by the primary investigator will be excluded from the study.
* Patients previously diagnosed with rheumatoid arthritis will be excluded from the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at their office visit scheduled with the principal investigator. Prior to the office visit, one of the surgeons diagnosed the potential subject with knee osteoarthritis. They recommended proceeding with a particular knee injection based upon previous treatments and insurance authorization. The determination of which injection is administered is not being determined by the study need.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in visual analog score at 3 months | 3 months
  The primary endpoint is significant improvement in visual analog scores for corticosteroid vs viscosupplementation injections pre- and post-injections. VAS scores range from 0-10, 0 being no pain, 10 being the worst pain imaginable. The hypothesis is the injections will help reduce the participant's perception of pain, resulting in lower VAS scores.
  If the power size is valid, VAS will be compared between males/females.

CONTACTS AND LOCATIONS:
Overall Officials: William J Vascik, MPAS, PA-C, Study Chair — Senior Physician Assistant
Locations (1):
- Three Rivers Orthopedic Associates, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No